CLINICAL TRIAL: NCT06174090
Title: The Effect of Patient Education With Video Prior to Coronary Artery Bypass Graft Surgery on Pain, Anxiety and Knowledge Levels of Patients
Brief Title: The Effect of Video Education on Pain, Anxiety and Knowledge Levels of Coronary Bypass Graft Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Gulcin Sahin, RN, MSc, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KA21/131
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: The intervention group will watch a 12-minute video-education about pre-post surgical process and care in bypass surgery, for once the day before surgery. Video-education was created by the researcher based on the literature. Expert opinion was provided related to content. The control group will receive standard verbal education lasting 12-minute about the issue.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-education (Experimental): Participants will receive video-education about bypass surgery care, the day before the surgery, for once.
  Interventions: Other: Coronary bypass graft surgery video education
- Control (No Intervention): Participants will receive verbal education about bypass surgery care, the day before the surgery, once

INTERVENTIONS:
Other: Coronary bypass graft surgery video education — It includes information about surgical process and handling issues within the first few days of surgery.
  Arms: Video-education

SUMMARY:
The aim of this research to examine the effectiveness of video-education on pain, anxiety, and knowledge levels on adult patients undergoing coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
A video based patient education will be used in this randomized controlled study. Patient education via video aims to reduce the patient's anxiety levels, control their pain, and improve their health outcomes by increasing knowledge levels. In addition, since this training is visual-based, it is aimed to provide effective learning by reducing the inequality due to sociodemographic and individual differences between participants. The video-education includes information about pre and post-surgical process and care.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* Being hospitalized in Cardiovascular Surgery Clinic and Cardiovascular surgery intensive care unit
* Undergoing coronary artery bypass graft surgery for the first time, by sternotomy method
* Patients who agree to participate in the research and read and sign the "Informed Volunteer Consent Form for Scientific Research"

Exclusion Criteria:

* Patients with visual or hearing impariment
* Patients with psychiatric illness,
* Patients with known cognitive impairment (dementia, Alzheimer's).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain Level | from 24th of surgery to 72nd hour
  Visual analog scale (VAS): VAS is a widely used scale for pain assessment. The scale was developed by Albersnagel, and its validity and reliability in our country were established by Aydin et al. In VAS, pain averages ranging from 0 to 10 are given on a 10 cm scale. Accordingly, while "0" indicates no pain, an average VAS value of "1-4" indicates mild pain, "5-6" indicates moderate pain, and "7-10" indicates severe. Change= VAS score of video-education group<standard verbal education.on 24th, 48th, and 72nd hours after surgery
Anxiety level | from baseline prior to education to 72nd hour of surgery
  State anxiety scale (STAI-I): The scale determines how the individual feels at a certain moment, in a certain condition, and his/her emotions regarding the situation. The total score obtained from the scale is between 20-80. A high score indicates a high level of anxiety. The feelings and behaviors expressed in the State Anxiety Scale items are answered by marking one of the following conditions, such as (1) not at all, (2) a little, (3) a lot and (4) completely, according to the severity of such experiences. Change= STAI-I score of video-education group<standard verbal education.on pre-and-post education, and on 72nd hours after surgery.
Preoperative anxiety | from baseline prior to education to 72nd hour of surgery
  Amsterdam Preoperative Anxiety and Information Scale (APAIS): The scale is one of the scales used to evaluate preoperative anxiety. Source of anxiety; It is divided into three: due to surgery, anesthesia or lack of information. It contains 6 statements regarding these three sources to assess anxiety. In order to objectify the survey, each statement is given a numerical value based on a 5-point Likert scale according to severity; These values, ranging from 1 to 5; 1=none, 2=mild, 3=moderate, 4=severe, 5=extreme severity. Higher score means higher preoperative anxiety. Change= APAIS score of video-education group<standard verbal education n pre-and-post education, and on 72nd hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Faculty of Health Sciences, Ankara, Etimesgut, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan for sharing IPD unless it is requested for a reasonable cause.